CLINICAL TRIAL: NCT02548260
Title: Treatment of Proximal Interphalangeal Joint Injuries. Comparative Study of the Clinical Efficiency and Cost of Syndactyly Treatment Versus Immobilization and Compression Versus no Compression
Brief Title: Treatment of Proximal Interphalangeal Joint Injuries. Clinical Efficiency of Syndactyly Treatment and Digital Compression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Thierry Christen, Staff physician, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 301/15
Record Dates: First submitted 2015-09-03; First posted 2015-09-14 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Finger Injuries
MeSH Terms: conditions — Finger Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Syndactyly without compression (Experimental): Relative immobilization with a syndactyly (CE conformity), no compression is worn.
  Interventions: Device: Syndactyly without compression
- Syndactyly with compression (Experimental): Relative immobilization with a syndactyly (CE conformity), compression (CE conformity) is worn over the finger
  Interventions: Device: Syndactyly with compression
- Rigid splint without compression (Experimental): Rigid immobilization with a custom made thermoplastic splint (CE conformity), no compression is worn
  Interventions: Device: Rigid splint without compression
- Rigid splint with compression (Experimental): Rigid immobilization with a custom made thermoplastic splint (CE conformity), compression (CE conformity) is worn over the finger
  Interventions: Device: Rigid splint with compression

INTERVENTIONS:
Device: Syndactyly without compression — three week relative immobilization by syndactyly
  Arms: Syndactyly without compression
Device: Syndactyly with compression — three week relative immobilization by syndactyly and compression
  Arms: Syndactyly with compression
Device: Rigid splint without compression — three week rigid immobilization by splint
  Arms: Rigid splint without compression
Device: Rigid splint with compression — three week rigid immobilization by splint and compression
  Arms: Rigid splint with compression

SUMMARY:
Proximal interphalangeal joint injuries of the fingers may be treated in various ways and no treatment has been shown to be superior. The investigators wish to study the effectiveness of syndactyly versus digital splint when comparing joint mobility. The investigators also wish to study the effectiveness of finger compression in reducing edema and therefore allowing a greater arc of motion.

DETAILED DESCRIPTION:
Proximal interphalangeal joint (PIPJ) injuries of the fingers are a common occurrence. They may be treated various ways: strict immobilization in a finger splint for one to three weeks, syndactyly, no immobilization. Immobilization is often responsible for joint stiffness whereas immediate mobilization might produce pain.

Injuries to the joints of the hand produce edema that is responsible for additional stiffness. Compressive garment may be worn to limit the extent of the edema and help its resorption.

Although PIPJ injuries are frequent, their treatment does not benefit from a consensus. Most studies are retrospective or aimed at a pediatric population. The investigators wish to evaluate the outcome of PIPJ injury after different treatments: either strict immobilization in a rigid splint for three weeks, of relative immobilization in a syndactyly for three weeks.The investigators also wish to study the effect of finger compression on edema resolution and finger motion. Therefore there will be four treatment groups: syndactyly with and without compression, rigid splint with and without compression.

The study will be conducted in the hand surgery unit of a university hospital in a prospective way. The assignment to a particular treatment group will be randomly performed. Patients will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* proximal interphalangeal joint injury with or without dorsal or lateral luxation
* less than seven days after injury
* injured joint stability
* fracture of the palmar rim of the intermediate phalanx less than 30% of articular surface

Exclusion Criteria:

* palmar luxation of the proximal interphalangeal joint
* fracture of the palmar rim of the intermediate phalanx greater than 30% of articular surface
* injury to the central band of the extensor tendon
* fracture other than palmar rim of the intermediate phalanx less than 30% of articular surface
* non reducible luxation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in digital mobility of wounded finger | 3 weeks, 6 weeks, 3 months, 6 months
  Evaluation of digital mobility by measuring the palm-tip of the finger distance with a ruler. The active and passive mobility of the metacarpophalangeal, proximal and distal interphalangeal joints will be measured with a goniometer.

SECONDARY OUTCOMES:
Change in pain | 3 weeks, 6 weeks, 3 months, 6 months
  Patient has to rate the pain in the wounded finger during the last two days using a visual analog scale.
Global function | 3 months
  Patient has to fill out the validated QuickDASH questionnaire relative to activities of daily living.
Satisfaction | 3 months
  Patient has to rate its satisfaction with the treatment outcome on a scale from 1 to 10 (greatest satisfaction = 10)
Cost | six months
  The cost of the whole treatment will be calculated for each patient after the final consultation at 6 months. It will include the consultations themselves, the cost of the devices used, the hand therapy, the absence from work.
Change in strength | 3 weeks, 6 weeks, 3 months, 6 months
  Pinch strength and global hand strength will be evaluated with specific devices (pinch and dynamometer)
Change in finger diameter | 3 weeks, 6 weeks, 3 months, 6 months
  Diameter of the injured finger at the proximal interphalangeal joint will be assessed with a specific device (rings of various diameter)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland